

# Participation in the trial of telehealth

This Statement is for your consent to participate in a trial of medical distance follow-up. The purpose of the trial is to find out how telehealth affects health, experience of the health service and consumption of health services. Participation is voluntary. You can withdraw your consent at any time. Below you can read more about the trial and what participation means to you and give your consent if you accept the invitation to participate.

#### What does participation mean to you?

- As a participant in the trial, you will be asked to complete a short questionnaire up to four times over 18 months, regardless of whether you are part of the group that receives follow-up using telehealth solutions or the control group. Your questionnaire responses are recorded electronically or on paper. In addition, some users will be asked to be interviewed by the researchers. It will take approximately one hour, and audio recordings and notes will be taken from the interviews.
- We will collect and record information about you from various local and national registers. All data will be de-identified, and results will be presented at group level. This means that you will not be able to recognize data that is being analyzed or presented. Table 1 (p. 4) gives an overview of what types of information are collected about you and from which registers.
- The purpose of the data collection is to investigate whether your state of health, experience and use of health services has changed during the trial period. This knowledge will help to further develop and improve the Norwegian health service.

## More about the testing

The Directorate of Health has been commissioned by the Ministry of Health and Care Services to

conduct a trial of medical distance monitoring in the period 2018-2021. The University of Oslo, Oslo Economics and the National Center for District Medicine are responsible for the research.

In practice, distance monitoring means that you as a user answer health-related questions on a tablet and/or record measurements related to your health (e.g. blood pressure, blood sugar, oxygen measurement). The information is sent electronically to a follow-up service, where health professionals monitor the measurements and follow you up in accordance with a treatment plan that your GP has prepared in consultation with you. The equipment is easy to use, and you get training at startup.

The purpose of the trial is to find out how distance follow-up affects the physical and mental health of users, user experience and use of resources in the health service. We will also examine how the service is delivered, and assess the costs and benefits of distance follow-up, both for the users, the health service and society as a whole. The Directorate of Health will

Notat, 8. august 2019



use the results of the research as the basis for national recommendations on distance followup.

In order to establish knowledge about the effect of distance follow-up compared to current practice, the test is conducted as a randomized controlled trial in selected municipalities. This means that half of those who agree to participate in the trial receive distance follow-up (so-called 'action group') while the other half receive regular follow-up from the health service (so-called 'control group'). It is a coincidence which group you end up in (is determined by lottery). To investigate the effect of distance monitoring on participants' consumption of health services in both the short and long term, we will collect and record information about you from various local and national registries in the period from 2017 to 2022. If your municipality continues the offer with distance follow-up after the end of the follow-up period (18 months), participants in both the action and control group will have the opportunity

### What happens to the information about you?

to be considered for distance follow-up.

The information recorded about you will be used as described above. You have the right to access the information that is registered about you and the right to correct any errors in the information that is registered. All information will be processed without name and birth number or any other directly recognizable information. A code links you to your information through a link key. Information obtained is stored on a secure data server. Audio recordings are stored in a locked safe, and notes are stored in a workbook that only the research group has access to on the Oslo Economics network. The project is scheduled to end on 31 December 2024, and audio recordings and information collected will be deleted within three years of the end of the project (by 31 December 2027). Information recorded about you by the employees in your municipality can be used for internal quality assurance in the municipality.

### Your rights

As long as you can be identified in the data material, you are entitled to:

- insight into what personal information is registered about you,
- obtaining personal information about you,
- to delete personal information about you,
- obtain a copy of your personal data (data portability), and
- to submit a complaint to the Privacy Ombudsman or the Data Inspectorate regarding the processing of your personal data.

# Approval of the test

We process information about you based on your consent.

On behalf of the Department of Health and Society at UiO and Oslo Economics, NSD - Norwegian Center for Research Data AS has considered that the processing of personal data in this project complies with the privacy regulations.



Voluntary participation and opportunity to consent

Participation in the trial is voluntary. If you wish to participate, sign the Declaration of Consent at the bottom of this page. You may withdraw your consent at any time and without giving any reason and may require that information collected about you be deleted. This will not have any impact on your continued use of the public health services. If you later want to retire or have questions about the project, you can contact:

Susanna Sten-Gahmberg, project manager at Oslo Economics, on mobile:

451 34 135, or by e-mail: ssg@osloeconomics.no. Alternatively, you can contact the Privacy Ombudsman at UiO by email: personvernombud@uio.no.

With best regards,

Tor Iversen Project Manager Professor at UiO

#### Consent Statement

I have received and understood information about the project Proof of medical distance follow-up and have been given the opportunity to ask questions. I agree to:

| Obtaining register information about me as described above (compulsory for |
|---|
| participation in the trial) |
| To participate in a survey (compulsory for participation in the test) |
| To participate in an interview |
| That my personal data is stored after the end of the project for research purposes |
| That my relatives can be interviewed about my participation in the trial |

I agree that my information will be processed until the project is completed and will be deleted by 31 December 2027.

(Signed by participant, date)

Table 1: Overview of information obtained from local and national registers

| Type opplysninger | Variabler | Kilde |
|---|---|---|
| General information about you | Age, gender, education, marital status, living situation and place of residence, main source of living (own income, pension, social security, other), household income (at intervals), extent of informal care, use of other types of welfare technology (security alarm, self-help tools, etc.) | Municipal registration and questionnaire |
| Your use of the GP services | Number of consultations and contacts, selected tariffs and measurements, number of kroner in the form of reimbursement and free cards | The Norwegian Health Economics Administration Database (KUHR), Municipal Patient and User Register (CPR), General practitioner register |
| Your use of the emergency room service, appointment specialists and physiotherapists with an operating agreement | Number of consultations and contacts, selected tariffs and measurements, number of kroner in the form of reimbursement and free cards | The Norwegian Health Economics Administration Database (KUHR), Municipal Patient and User Register (KPR) |
| Your use of municipal health and care services | Number of visits and time spent on home services and practical assistance, municipal emergency 24-hour service, short-term stays | Municipal Patient and<br>User Register (KPR),<br>electronic patient<br>record |
| Your use of specialist health services | Information on outpatient consultations, bed days, admissions including procedures and diagnoses | Norwegian Patient<br>Register (NPR) |
| Your use of telehealth | Date of start-up and eventual termination, recruitment channel, status, diagnoses, assigned technology | Municipal registration |
| Your measurements<br>and other records from<br>the follow-up service | Answers to questions about your health, measurements of weight, blood sugar, blood pressure, oxygen measurement, heart rate, spirometry, temperature and other measurements from the test | Follow-up service / municipality / technical solution provider |
| Your use of medicines | Use of medicines; number, types and doses | Norwegian<br>Prescription Database<br>(NorPD) |

Notat, 8. august 2019